CLINICAL TRIAL: NCT02636491
Title: Open-label, 3 Center, Randomized, Cross-over Study to Evaluate the Safety and Efficacy of 60 Hours Closed-loop Control Using the MD-Logic Automated Insulin Delivery System Compared to Sensor Augmented Pump Therapy at T1D Patients at Home
Brief Title: Use of an Automated Insulin Delivery System Compared to Sensor Augmented Pump at Patients With Type 1 Diabetes (T1D)
Acronym: DREAM5
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kinderkrankenhaus auf der Bult (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MC-01
Record Dates: First submitted 2015-12-17; First posted 2015-12-21 (Estimated); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- investigational device (Experimental): MD-Logic-Automated Insulin Delivery System, Version 01.05.02
  The device is being used continuously over 60 hours for insulin therapy
  Interventions: Device: MD-Logic-Automated Insulin Delivery System
- MiniMed Paradigm® Veo™ System (Placebo Comparator): sensor augmented insulin pump
  The device is being used continuously over 60 hours for insulin therapy
  Interventions: Device: MiniMed Paradigm® Veo™ System

INTERVENTIONS:
Device: MD-Logic-Automated Insulin Delivery System — Subjects will undergo 60 hours at home under MD-Logic control and continuing with their regular routine life. At evening of the first intervention day patients will switch to MD-Logic control. Patients will be asked to connect study sensor and pump to the computer using the MD-Logic software. After the activation of the MD-Logic system, basal insulin dosing and correction boluses will be fully automated and controlled by the MD-Logic system except to meal boluses. Patients will be encouraged to measure capillary blood glucose at least 4 times a day, before each meal and before bed time. After the third night the patient will turn the closed-loop controller "OFF", this will automatically save the log file. The patient will return to his regular insulin treatment.
  Other Names: Closed loop
  Arms: investigational device
Device: MiniMed Paradigm® Veo™ System — Subjects use 60 hours at home their conventional insulin pump and continuing with their regular Routine life. During this therapy the Insulin pump operating separately and are not controlled by the MD-Logic System.
  Other Names: sensor augmented continuous subcutaneous insulin infusion
  Arms: MiniMed Paradigm® Veo™ System

SUMMARY:
Title: An open-label, three-center, randomized, cross-over study to evaluate the safety and efficacy of day and night closed-loop control using the MD-Logic automated insulin delivery system compared to sensor augmented pump therapy at patients with type 1 diabetes at home Indication: Type 1 Diabetes mellitus using an insulin pump therapy and continues glucose sensors The objective of this pilot study is to evaluate the safety and efficacy of 60 hours blood glucose control, using the MD-Logic System in individuals with type 1 diabetes at patient's home.

The duration of study participation for one subject is 28-56 days and the overall duration of the study is 6 months The participants of the study are patients ≥ 10 years until 65 years with Type 1 Diabetes mellitus using and insulin pump therapy and continuous glucose sensors.

Sample Size n = 45

DETAILED DESCRIPTION:
Up to 45 eligible patients will be enrolled to participate in two crossover sessions of 60 hours of consecutive days, with closed-loop or sensor-augmented pump therapy (Minimed ®Paradigm). The sequence of the sessions will be randomly assigned. The randomization will be blocked randomization (1:1). Patients will be assigned to one of the following arm: Group A: 60 hours under closed-loop control and then 60 hours of sensor augmented pump therapy and Group B: 60 hours using sensor augmented pump therapy and then 60 hours under closed-loop control.

Subjects will be enrolled according to the following schedule/ successive phases:

Phase 1: 5 Adult subjects: After all adult subjects have completed the study the 2nd enrollment phase starts.

Phase 2: 5 Adolescent subjects aged 14-18. After these subjects have completed the study the 3rd enrollment phase starts.

Phase 3: 5 Children aged 10-14 will be enrolled.

The enrollment of phase 2 and phase 3 will not be started before all participants of the previous phase completed the study and the safety and efficacy of the system has been analyzed based on the occurrence of (serious) adverse Events (AE) or any other issue relevant for patient's safety. If the observed AEs or device problems do not exceed the amount or severity of the risks expected during a regular diabetes therapy and the recruitment of the next age category is considered reasonable from the medical point of view, the next enrollment phase will be started.Screening Failures will be replaced to get a total of 45 completed patients.The average duration of study participation for subjects completing the study is estimated to be approximately 28-56 days. The estimated duration of the total study is 6 months.In this study 45 patients will be included, 15 are planned to be enrolled in Germany.

The study will consist of 5 visits (3 clinical visits and 2 visits will be done by phone) as followed:

* Visit 1: Screening, eligibility, enrolment and sensor and diabetes guidelines training. (Day - 21)
* Run-in period
* Visit 2: Randomization and preparation visit for the outpatient period. (Day 0)
* Intervention session 1 (same weekdays as Intervention session 2)
* Visit 3: Phone call visit between arms. (Day 4)
* Washout period
* Visit 4: Phone call visit before session 2 (Day 18)
* Intervention session 2 (same weekdays as Intervention session 1)
* Visit 5: Final visit. (Day 21)

There is no follow up visit or observation planned after the end of the study or after a subject discontinued study participation. In case of a Serious Adverse Event (SAE) a follow up period until this SAE is resolved/ recovered is planned.

ELIGIBILITY:
Inclusion Criteria:

1. Subject with Type 1 diabetes (>1yr since diagnosis)
2. Insulin infusion pump (CSII) therapy for at least 3 months
3. Patients using a Continuous glucose monitoring system
4. Age ≥ 10 years until 65 years
5. HbA1c at inclusion ≥ 7 and <10
6. Patients willing to follow study instructions
7. Patients live with at least one other adult person
8. BMI SDS (Standard Deviation Scores) - below the 95th percentile for age32
9. Patients with care givers who are capable of operating a computer based system.

Exclusion Criteria:

1. Concomitant diseases that influence metabolic control (e.g. anemia, significantly impaired hepatic function, renal failure, History of adrenal insufficiency) or other medical condition, which in the Investigator's opinion, may compromise patient safety as the following examples:

   * Abnormal liver or renal function (Transaminase >2 times the upper limit of normal, Creatinine > 1.5 mg/dL)
   * Subject has had any of the following diagnoses within 1 year of screening: myocardial infarction, unstable angina, coronary artery disease or congestive heart failure, coronary artery surgery, transient ischemic attack, cerebrovascular accident, uncontrolled hypertension, ventricular rhythm disturbances or thromboembolic disease Note: Adequately treated thyroid disease and celiac disease do not exclude subjects from enrollment
2. Participation in any other interventional study
3. Known or suspected allergy to trial products such as adhesives, tapes, needles. An allergy to contrast medium, use of other active medical devices (such as pacemaker, ICD) and planned imaging examinations (such as MRI).
4. Any significant diseases or conditions including psychiatric disorders and substance abuse that, in the opinion of the investigator, is likely to affect the subject's ability to complete the study, or compromise patient safety
5. Diabetic ketoacidosis in the past 1 month.
6. Severe hypoglycemia six month prior to enrollment.
7. Current use of the following medications: medications that are used to lower blood glucose such as Pramilintide, Metformin and GLP-1 (Glucagon-like Peptide-1) analogs. Beta blockers, glucocorticoids and other medications, which in the judgment of the investigator would be a contraindication to participation in the study
8. Subject is participating in another drug or device study that could affect glucose measurements or glucose management.
9. Female subject who is pregnant or breast-feeding or is planning to become pregnant within the planned study duration.
10. Not sufficient vision or hearing to recognize pump/ sensor alarms or to perform blood glucose -self measurements 4-times daily.
11. Relevant severe organ disorders (diabetic nephropathy, diabetic retinopathy, , diabetic foot syndrome) or any secondary disease or complication of diabetes mellitus

    * Subject has unstable or rapidly progressive renal disease or is receiving dialysis
    * Subject has active proliferating retinopathy
    * Active gastroparesis
12. Patient suffers from an eating disorder

Ages: 10 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2015-12; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
normal glucose level | 60 hours
  Percentage of Glucose sensor readings within 70 to 180mg/dl (3.9 to 10 mmol/l)

SECONDARY OUTCOMES:
Hypoglycemia | 60 hours
  Percentage of glucose sensor readings below 70 mg/dl (3.9 mmol/l)
increased glucose level | 60 hours
  Percentage of glucose sensor readings above 180mg/dl (10 mmol/l)
glucose sensor readings | 90 hours
  Average and Standard deviation of glucose sensor readings

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Danne, MD, Principal Investigator — Kinder- und Jugendkrankenhaus AUF DER BULT
Locations (1):
- Kinder - und Jugendkrankenhaus AUF DER BULT, Hanover, Germany

IPD SHARING:
Plan to Share IPD: No